CLINICAL TRIAL: NCT04368429
Title: Immunogenicity and Safety of a Single Dose of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Children, Adolescents, and Adults 2 to 55 Years of Age
Brief Title: Study of a Quadrivalent Meningococcal Conjugate Vaccine as a Single Dose Compared With a Single Dose of a Meningococcal Reference Vaccine in Children, Adolescents, and Adults 2 to 55 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EFC16335; MEQ00068 (UTN); U1111-1241-8382 (Other: UTN)
Record Dates: First submitted 2020-04-20; First posted 2020-04-29 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Meningococcal Immunisation (Healthy Volunteers)
MeSH Terms: interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: MenACYW Conjugate Vaccine (Experimental): Participants received a single intramuscular (IM) dose of MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine (MenACYW Conjugate Vaccine)
- Group 2: Menactra® vaccine (Active Comparator): Participants received a single IM dose of Menactra® vaccine on Day 0.
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine (MenACYW Conjugate Vaccine) — Pharmaceutical form: Liquid solution Route of administration: IM
  Arms: Group 1: MenACYW Conjugate Vaccine
Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — Pharmaceutical form: Liquid solution Route of administration: IM
  Other Names: Menactra®
  Arms: Group 2: Menactra® vaccine

SUMMARY:
Primary Objective:

To demonstrate the non-inferiority of the antibody responses to meningococcal serogroups A, C, Y, and W following the administration of a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine (MenACYW Conjugate vaccine) compared with those observed following the administration of a single dose of Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra® vaccine).

Secondary Objective:

Immunogenicity: To describe the antibody responses to the meningococcal serogroups A, C, Y, and W before and 30 days (+14 days) after vaccination with MenACYW Conjugate vaccine or Menactra®.

Safety: To describe the safety profile of MenACYW Conjugate vaccine and that of Menactra®.

DETAILED DESCRIPTION:
The duration of each participant's participation in the study was approximately 30 to 44 days.

ELIGIBILITY:
Inclusion criteria :

* Aged 2 to 55 years on the day of inclusion.
* Informed consent form had been signed and dated by the participants or participants' parents/legally acceptable representatives as applicable. In addition: Participants 7 to 19 years provided written assent.
* Participants (and participants' parents/legally acceptable representatives for the 2 to 19 years age groups) were able to attend all scheduled visits and complied with all study procedures.

Exclusion criteria:

* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception* or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination).

  *Effective methods of contraception included oral contraception (pill), intrauterine device, or condoms used with spermicide.
* Participation in the 4 weeks preceding the study vaccination or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine prior to Visit 2 except for influenza vaccination, which may be received at least 2 weeks before or after the study investigational vaccines. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal disease with either the study vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or Conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B vaccine).
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the study (specifically, but not limited to, subjects with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances.
* Laboratory confirmed / self-reported thrombocytopenia, contraindicating IM vaccination in the Investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination in the Investigator's judgement.
* History of Guillain-Barre syndrome.
* History of convulsions.
* History of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine and a diphtheria toxoid-containing vaccine within 10 years of the proposed study vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature greater than or equal to (>=) 99.5 degree Fahrenheit or >= 37.5 degree Celsius). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2020-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- Japan (4):
  - Investigational Site Number 3920001, Koganeishi
  - Investigational Site Number 3920004, Nagoya
  - Investigational Site Number 3920002, Shinjuku-Ku
  - Investigational Site Number 3920003, Shinjuku-Ku

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC16335 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25245&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled at 4 active centers in Japan from 22 May 2020 to 05 October 2020.
Pre-assignment Details: A total of 360 participants were enrolled and randomized in the study.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Participants received a single intramuscular (IM) dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate vaccine (MenACYW Conjugate vaccine) on Day 0.
- Group 2: Menactra® Vaccine: Participants received a single IM dose of Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra® vaccine) on Day 0.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Started | 180 | 180
Safety Analysis Set (Participants who received at least one dose of the study vaccine and had any safety data available; analyzed according to the vaccine they actually received.) | 179 | 180
Completed | 179 | 180
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Participants received a single IM dose of MenACYW Conjugate vaccine on Day 0.
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine | Total
Number analyzed (Participants) | 180 | 180 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (11.09) | 24.1 (10.27) | 24.6 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 95 | 179
  Male | 96 | 85 | 181
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 180 | 180 | 360
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Vaccine Seroresponse For Meningococcal Serogroup A, C, Y And W Following Vaccination With MenACYW Conjugate and Menactra® Vaccine: Non-Inferiority Analysis
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by serum bactericidal assay using human complement (hSBA). The hSBA vaccine seroresponse was defined as a post-vaccination hSBA titer greater than or equal to (>=) 1:16 for participants with pre-vaccination hSBA titer less than (<) 1:8, or a >= 4-fold increase in hSBA titer from pre-vaccination to post-vaccination for participants with pre-vaccination hSBA titer >= 1:8.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on Per-Protocol Analysis Set (PPAS) population that included participants who received 1 dose of the study vaccine and had a valid post-vaccination blood sample result with no relevant protocol deviations. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Number analyzed (Participants) | 174 | 179
percentage of participants
  Serogroup A | 85.6 [79.5 to 90.5] | 65.4 [57.9 to 72.3]
  Serogroup C | 96.6 [92.6 to 98.7] | 62.6 [55.0 to 69.7]
  Serogroup Y: number analyzed (Participants) | 174 | 178
  Serogroup Y | 97.7 [94.2 to 99.4] | 63.5 [56.0 to 70.6]
  Serogroup W | 87.4 [81.5 to 91.9] | 49.2 [41.6 to 56.7]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menactra® Vaccine; Serogroup A; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% Confidence Interval (CI) of the difference in percentage was greater than (>) -10% for the serogroup A; Difference in percentage = 20.27, 95% CI 2-sided [11.38 to 28.75] — 95% CI of the difference in percentage was calculated from the Wilson Score method without continuity correction
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menactra® Vaccine; Serogroup C; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference in percentage was >-10% for the serogroup C; Difference in percentage = 33.98, 95% CI 2-sided [26.20 to 41.50] — 95% CI of the difference in percentage was calculated from the Wilson Score method without continuity correction
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menactra® Vaccine; Serogroup Y; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference in percentage was >-10% for the serogroup Y; Difference in percentage = 34.22, 95% CI 2-sided [26.66 to 41.64] — 95% CI of the difference in percentage was calculated from the Wilson Score method without continuity correction
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menactra® Vaccine; Serogroup W; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference in percentage was >-10% for the serogroup W; Difference in percentage = 38.19, 95% CI 2-sided [28.93 to 46.53] — 95% CI of the difference in percentage was calculated from the Wilson Score method without continuity correction

2. Secondary Outcome: Percentage of Participants With Vaccine Seroresponse For Meningococcal Serogroup A, C, Y And W Following Vaccination With MenACYW Conjugate and Menactra® Vaccine
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. The hSBA vaccine seroresponse was defined as a post-vaccination hSBA titer >=1:16 for participants with pre-vaccination hSBA titer <1:8, or a >= 4-fold increase in hSBA titer from pre-vaccination to post-vaccination for participants with pre-vaccination hSBA titer >= 1:8.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS population. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Number analyzed (Participants) | 174 | 179
percentage of participants
  Serogroup A | 85.6 [79.5 to 90.5] | 65.4 [57.9 to 72.3]
  Serogroup C | 96.6 [92.6 to 98.7] | 62.6 [55.0 to 69.7]
  Serogroup Y: number analyzed (Participants) | 174 | 178
  Serogroup Y | 97.7 [94.2 to 99.4] | 63.5 [56.0 to 70.6]
  Serogroup W | 87.4 [81.5 to 91.9] | 49.2 [41.6 to 56.7]

3. Secondary Outcome: Percentage of Participants With hSBA Antibody Titer >=1:4 and >=1:8 Following Vaccination With MenACYW Conjugate and Menactra® Vaccine
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. Percentage of participants With hSBA antibody titers >=1:4 and >=1:8 for serogroups A, C, Y, and W were reported in the outcome measure.
Time Frame: Day 0 (pre-vaccination); Day 30 (post-vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Number analyzed (Participants) | 174 | 179
percentage of participants
  Serogroup A: >= 1:4: Day 0 | 82.8 [76.3 to 88.1] | 82.1 [75.7 to 87.4]
  Serogroup A: >= 1:8: Day 0 | 42.5 [35.1 to 50.2] | 46.9 [39.4 to 54.5]
  Serogroup A: >= 1:4: Day 30 | 98.3 [95.0 to 99.6] | 98.9 [96.0 to 99.9]
  Serogroup A: >= 1:8: Day 30 | 96.6 [92.6 to 98.7] | 92.7 [87.9 to 96.1]
  Serogroup C: >= 1:4: Day 0 | 55.2 [47.5 to 62.7] | 65.9 [58.5 to 72.8]
  Serogroup C: >= 1:8: Day 0 | 31.6 [24.8 to 39.1] | 38.5 [31.4 to 46.1]
  Serogroup C: >= 1:4: Day 30 | 100 [97.9 to 100] | 90.5 [85.2 to 94.4]
  Serogroup C: >= 1:8: Day 30 | 98.9 [95.9 to 99.9] | 81.0 [74.5 to 86.5]
  Serogroup Y: >= 1:4: Day 0: number analyzed (Participants) | 174 | 178
  Serogroup Y: >= 1:4: Day 0 | 39.7 [32.3 to 47.3] | 44.9 [37.5 to 52.6]
  Serogroup Y: >= 1:8: Day 0: number analyzed (Participants) | 174 | 178
  Serogroup Y: >= 1:8: Day 0 | 27.0 [20.6 to 34.3] | 29.2 [22.7 to 36.5]
  Serogroup Y: >= 1:4: Day 30 | 100 [97.9 to 100] | 97.2 [93.6 to 99.1]
  Serogroup Y: >= 1:8: Day 30 | 100 [97.9 to 100] | 89.4 [83.9 to 93.5]
  Serogroup W: >= 1:4: Day 0 | 73.0 [65.7 to 79.4] | 76.0 [69.0 to 82.0]
  Serogroup W: >= 1:8: Day 0 | 51.1 [43.5 to 58.8] | 58.7 [51.1 to 66.0]
  Serogroup W: >= 1:4: Day 30 | 100 [97.9 to 100] | 96.6 [92.8 to 98.8]
  Serogroup W: >= 1:8: Day 30 | 99.4 [96.8 to 100] | 91.1 [85.9 to 94.8]

4. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroup A, C, Y And W Following Vaccination With MenACYW Conjugate and Menactra® Vaccine
Description: GMTs of antibodies against meningococcal serogroups A, C, Y, and W were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 0 (pre-vaccination); Day 30 (post-vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Number analyzed (Participants) | 174 | 179
titers
  Serogroup A: Day 0 | 5.79 [5.06 to 6.63] | 5.96 [5.28 to 6.73]
  Serogroup A: Day 30 | 123 [99.4 to 152] | 41.3 [33.3 to 51.3]
  Serogroup C: Day 0 | 4.47 [3.86 to 5.18] | 5.27 [4.53 to 6.12]
  Serogroup C: Day 30 | 544 [431 to 685] | 36.6 [28.3 to 47.5]
  Serogroup Y: Day 0: number analyzed (Participants) | 174 | 178
  Serogroup Y: Day 0 | 3.95 [3.36 to 4.65] | 4.29 [3.62 to 5.08]
  Serogroup Y: Day 30 | 221 [183 to 267] | 41.5 [32.7 to 52.6]
  Serogroup W: Day 0 | 7.39 [6.21 to 8.79] | 8.41 [7.09 to 9.98]
  Serogroup W: Day 30 | 125 [104 to 151] | 36.5 [29.3 to 45.5]

5. Secondary Outcome: Percentage of Participants With hSBA Titers Following Vaccination With MenACYW Conjugate and Menactra® Vaccine
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA. Percentage of participants with hSBA titers <1:4, 1:4, 1:8, 1:16,1:32, 1:64, 1:128, 1:256, 1:512, 1:1024, 1:2048 and 1:4096 for serogroups A, C, Y, and W; with hSBA titers of 1:8192 for serogroup Y; and with hSBA titers of 1:8192, 1:16384, 1:32768 for serogroup C were reported.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Number analyzed (Participants) | 174 | 179
percentage of participants
  Serogroup A:<1:4 | 1.7 | 1.1
  Serogroup A: 1:4 | 1.7 | 6.1
  Serogroup A: 1:8 | 2.9 | 12.3
  Serogroup A: 1:16 | 4.6 | 18.4
  Serogroup A: 1:32 | 11.5 | 17.9
  Serogroup A: 1:64 | 13.2 | 14.5
  Serogroup A: 1:128 | 24.1 | 13.4
  Serogroup A: 1:256 | 16.1 | 8.9
  Serogroup A: 1:512 | 15.5 | 2.8
  Serogroup A: 1:1024 | 7.5 | 3.9
  Serogroup A: 1:2048 | 0.6 | 0
  Serogroup A: 1:4096 | 0.6 | 0.6
  Serogroup C:<1:4 | 0 | 9.5
  Serogroup C: 1:4 | 1.1 | 9.5
  Serogroup C: 1:8 | 0.6 | 8.9
  Serogroup C: 1:16 | 2.3 | 10.1
  Serogroup C: 1:32 | 3.4 | 15.1
  Serogroup C: 1:64 | 4.0 | 14.0
  Serogroup C: 1:128 | 7.5 | 14.5
  Serogroup C: 1:256 | 12.6 | 8.4
  Serogroup C: 1:512 | 22.4 | 5.6
  Serogroup C: 1:1024 | 25.9 | 3.9
  Serogroup C: 1:2048 | 8.6 | 0
  Serogroup C: 1:4096 | 7.5 | 0.6
  Serogroup C: 1:8192 | 1.7 | 0
  Serogroup C: 1:16384 | 1.1 | 0
  Serogroup C: 1:32768 | 1.1 | 0
  Serogroup Y:<1:4 | 0 | 2.8
  Serogroup Y:1:4 | 0 | 7.8
  Serogroup Y:1:8 | 0.6 | 11.7
  Serogroup Y: 1:16 | 1.7 | 15.1
  Serogroup Y: 1:32 | 6.9 | 16.8
  Serogroup Y: 1:64 | 16.1 | 19.0
  Serogroup Y: 1:128 | 20.7 | 7.8
  Serogroup Y: 1:256 | 20.7 | 6.1
  Serogroup Y: 1:512 | 14.4 | 8.4
  Serogroup Y: 1:1024 | 12.6 | 2.8
  Serogroup Y: 1:2048 | 4.0 | 1.7
  Serogroup Y: 1:4096 | 1.1 | 0
  Serogroup Y: 1:8192 | 1.1 | 0
  Serogroup W:<1:4 | 0 | 3.4
  Serogroup W:1:4 | 0.6 | 5.6
  Serogroup W:1:8 | 1.7 | 10.1
  Serogroup W:1:16 | 5.2 | 19.6
  Serogroup W:1:32 | 13.8 | 24.6
  Serogroup W:1:64 | 16.1 | 14.5
  Serogroup W:1:128 | 25.3 | 9.5
  Serogroup W:1:256 | 19.0 | 3.4
  Serogroup W:1:512 | 10.3 | 2.2
  Serogroup W:1:1024 | 6.3 | 7.3
  Serogroup W:1:2048 | 1.1 | 0
  Serogroup W:1:4096 | 0.6 | 0

6. Secondary Outcome: Percentage of Participants With >=4-Fold Rise In hSBA Titers Following Vaccination With MenACYW Conjugate and Menactra® Vaccine
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA.
Time Frame: From Baseline (Day 0) to Day 30 (post-vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Number analyzed (Participants) | 174 | 179
percentage of participants
  Serogroup A | 85.6 [79.5 to 90.5] | 65.4 [57.9 to 72.3]
  Serogroup C | 96.6 [92.6 to 98.7] | 62.6 [55.0 to 69.7]
  Serogroup Y: number analyzed (Participants) | 174 | 178
  Serogroup Y | 97.7 [94.2 to 99.4] | 63.5 [56.0 to 70.6]
  Serogroup W | 87.4 [81.5 to 91.9] | 49.2 [41.6 to 56.7]

7. Secondary Outcome: Number of Participants Reporting Immediate Adverse Events (AEs) Following Vaccination With MenACYW Conjugate and Menactra® Vaccine
Description: An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination. All participants were observed for 30 minutes after vaccination, and any unsolicited systemic AEs occurred during that time were recorded as immediate unsolicited AEs in the CRB.
Time Frame: Within 30 minutes post-vaccination
Population: Analysis was performed on Safety Analysis Set which included participants who received at least one dose of the study vaccine and had any safety data available; analyzed according to the vaccine they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Number analyzed (Participants) | 179 | 180
Participants | 0 | 0

8. Secondary Outcome: Number of Participants Reporting Solicited Injection Site And Systemic Reactions Following Vaccination With MenACYW Conjugate and Menactra® Vaccine
Description: A solicited reaction was an expected adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRB and considered as related to the administered vaccination. Solicited injection site reactions included pain, erythema, swelling, and induration. Solicited systemic reactions included fever, headache, malaise and myalgia.
Time Frame: Within 7 days post-vaccination
Population: Analysis was performed on Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Number analyzed (Participants) | 179 | 180
Participants
  Injection site pain | 72 | 66
  Injection site erythema | 16 | 8
  Injection site swelling | 14 | 6
  Injection site induration | 6 | 5
  Fever | 3 | 1
  Headache | 34 | 17
  Malaise | 22 | 9
  Myalgia | 38 | 30

9. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events Following Vaccination With MenACYW Conjugate and Menactra® Vaccine
Description: An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRB in terms of diagnosis and/or onset window post-vaccination.
Time Frame: Up to 30 days post-vaccination
Population: Analysis was performed on Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Number analyzed (Participants) | 179 | 180
Participants | 15 | 11

10. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) Following Vaccination With MenACYW Conjugate and Menactra® Vaccine
Description: An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event.
Time Frame: From Day 0 up to 30 days post-vaccination
Population: Analysis was performed on Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
Number analyzed (Participants) | 179 | 180
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AE data were collected from Day 0 (pre-vaccination) up to Day 30 (post-vaccination). Solicited reactions were collected within 7 days post-vaccination. Serious AEs data were collected throughout the trial (i.e., up to 30 days post-vaccination).
Description: Analysis was performed on Safety Analysis Set.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menactra® Vaccine
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/180
Serious Adverse Events (participants affected / at risk) | 0/179 | 0/180
Other Adverse Events (participants affected / at risk) | 98/179 | 83/180
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=179) | Group 2: Menactra® Vaccine (N=180)
Injection Site Erythema (General disorders) | 16 (16) | 8 (8)
Injection Site Pain (General disorders) | 72 (72) | 66 (66)
Injection Site Swelling (General disorders) | 14 (14) | 6 (6)
Malaise (General disorders) | 22 (22) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 38 (38) | 30 (30)
Headache (Nervous system disorders) | 36 (36) | 17 (17) — Headache events that occurred after 7 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT04368429/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT04368429/SAP_001.pdf